CLINICAL TRIAL: NCT03931226
Title: Impact of Spa Treatments on the Consumption of Care in Children
Acronym: PEDIATHERM
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0420
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Respiratory Disease; Otorhinolaryngologic Diseases; Dermatologic Disease
Keywords: drug consumption
MeSH Terms: conditions — Respiration Disorders; Otorhinolaryngologic Diseases; Skin Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Departmental cohort: Department level of the Haute-Garonne through the use of the 'POMME' cohort (PrescriptiOns Medicines Mother Children)
  Interventions: Drug: Drug consumption
- National cohort: National level through the use of the "EGB" database (General Sample of Beneficiaries)
  Interventions: Drug: Drug consumption

INTERVENTIONS:
Drug: Drug consumption — number of Daily Defined Doses (DDDs) of medications prescribed and given to children in connection with the indication of the spa treatment

SUMMARY:
Children represent 1.2% of the spa population in France. Spa treatments, including climatic stays, are mainly prescribed for children in the context of respiratory, otorhinolaryngology and dermatological conditions. The benefits after spa treatments are the improvement of the symptoms of the pathology, the quality of life and in particular the reduction of drug exposures.

Few authors have recently investigated the impact of spa treatments on the health of children and society, while care has changed significantly in recent years. Moreover, no real-life study of a large sample of children seems to have been conducted in this area. The present study plan to conduct a pharmacoepidemiology study on medico-administrative databases of the "observational study" type, in real life.

ELIGIBILITY:
Inclusion Criteria:

* Children living in France at the time of the study
* 'POMME' cohort : children included at birth and 'EGB' cohort : children from birth to 15 years-old

Exclusion Criteria:

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This pharmacoepidemiology study of the "observational study" type, in real life, will concern children aged 1 to 15 living in France at the time of the study. It will be conducted at the departmental level of the Haute-Garonne through the use of the APPLE database (PrescriptiOns Medicines Mother Children) and at the national level through the use of the database. EGB (General Sample of Beneficiaries).
Sampling Method: Non-Probability Sample
Enrollment: 8372 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Drug consumption | until 7 years-old of children
  number of Daily Defined Doses (DDDs)

SECONDARY OUTCOMES:
Description of spa treatment | until 7 years-old of children
  Number and type of spa treatment
Population of children | until 7 years-old of children
  population of children in terms of age, weight and weight characteristics and health through compulsory health certificates at 8 days, 9 months and 2 years, but also use of care and medication
Compare 2 data sources | until 7 years-old of children
  Compare the population of children from the 2 data sources used for this project (departmental level with the cohort 'POMME' and national level with the 'EGB') to determine if the geographical situation of the department of Haute-Garonne influences the management of this type of diseases
impact of SPA treatment on the pathology | until 7 years-old of children
  Study the impact of spa treatments on the consumption of care in connection with the pathology that motivated the spa treatment, before and after the SPA
Medical costs | until 7 years-old of children
  impact of spa treatments on the consumption of medicines and care in terms of cost to society.

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Sommet, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No